CLINICAL TRIAL: NCT06114212
Title: Phase 1 Open-Label Pilot Trial of Deep Repetitive Transcranial Stimulation of the Lateral Prefrontal Cortex and Insula for Adults with Moderate-to-Severe Cannabis Use Disorder
Brief Title: Deep Repetitive Transcranial Magnetic Stimulation for Cannabis Use Disorder
Acronym: TRANS-CANN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, James MacKillop, Director, Peter Boris Centre for Addiction Research; Director, Michael G. DeGroote Centre for Medicinal Cannabis Research, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16698
Record Dates: First submitted 2023-10-06; First posted 2023-11-02 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Cannabis Use Disorder
Keywords: Transcranial Magnetic Stimulation; H4 coil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- H4 dTMS (Experimental): The participants will receive 18 H4 dTMS sessions over 4-6 weeks as an adjunct to evidence-based standard care for CUD (i.e., motivational interviewing and contingency management).
  Interventions: Device: dTMS stimulation via the H4 coil

INTERVENTIONS:
Device: dTMS stimulation via the H4 coil — Deep repetitive transcranial magnetic stimulation (dTMS) uses transient electromagnetic fields to stimulate the brain and is approved by Health Canada and the FDA for the treatment of depression, anxious depression, obsessive-compulsive disorder, and tobacco use disorder. Compared to the traditional TMS, dTMS is able to target brain depths ranging from 2 to 6 cm. With the use of various H-coils, dTMS has been used to target specific neural networks with the aim of producing desired clinical effects in psychiatric populations. The intervention in this study is the H4 dTMS coil which stimulates the lateral prefrontal cortex and the insula in the brain.

SUMMARY:
There is a credible basis for lateral prefrontal cortex and insula deep repetitive transcranial magnetic stimulation (dTMS) stimulation as a treatment for cannabis use disorder (CUD), but no studies to date have examined this. Evidence of benefit could expand the treatment options available for CUD but require randomized controlled trials (RCTs) to evaluate its efficacy. Toward an RCT of this intervention, the proposed study is a phase 1 open-label pilot trial of dTMS for adults with CUD. This study will establish the viability of an H4 protocol constituting an active arm of a future double-blind RCT.

DETAILED DESCRIPTION:
Deep repetitive transcranial magnetic stimulation (dTMS) is a technique that stimulates areas of the brain using magnetic pulses and is an approved treatment for several mental health and substance use disorders. The treatment uses head coils to deliver the magnetic pulses. A dTMS coil called the H4 coil stimulates the lateral prefrontal cortex and insula, and has been approved for the treatment of tobacco use disorder. No studies have been conducted on the H4 coil for treat cannabis use disorder. The purpose of this pilot study is to determine feasibility and tolerability of a dTMS H4 protocol. The goal is to lay the foundation for randomized controlled trials of dTMS as a treatment for adults with moderate-to-severe cannabis use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age 25-65
* DSM-5 CUD, moderate or higher (4+ DSM-5 symptoms)
* 4 or more days of cannabis use per week
* Reports inhalation as one route of administration
* Treatment-seeking (i.e., self-reported readiness to change of 5 or greater on a 0-10 readiness ruler)
* Stable domicile and reliable transportation, and willingness to attend in-person visits at SJHH Hamilton.

Exclusion Criteria:

* Current psychotic symptoms, history of schizophrenia-spectrum disorders or bipolar disorder, or current PTSD
* Active suicidality (past 3 months) or history of severe suicidality (i.e., requiring hospitalization)
* Any other mental health condition deemed incompatible by the team
* High risk alcohol involvement and/or 4+ symptoms of alcohol use disorder
* Unstable management of an existing mental health condition or anticipation of a change to the treatment over the next 3 months
* Current unstable medical condition (e.g., diabetes)
* rTMS Contraindications: intracranial or metal implants in the head or nearby regions that cannot be safely removed; history of epilepsy or seizures; pregnancy (female participants only); pacemaker and/or implantable cardioverter-defibrillators).
* Medication contraindications (e.g., bupropion >300 mg/day due to risk of seizures, benzodiazepine equivalent dose to lorazepam >2 mg/day).
* History of recurrent headache or migraine (past year)
* Significant literacy, visual, or hearing problems
* Co-enrollment in a clinical drug trial

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of H4 deep dTMS coils in adults with cannabis use disorder. | End of intervention period (~4 weeks)
  To determine the protocol feasibility, the percentage of intervention sessions completed by the participants will be examined
Tolerability of H4 deep dTMS coils in adults with cannabis use disorder. | End of intervention period (~4 weeks)
  To determine the protocol tolerability, the percentage of withdrawn participants will be examined
Safety of H4 deep dTMS coils in adults with cannabis use disorder. | End of intervention period (~4 weeks)
  To determine the protocol safety, weekly adverse events reported will be examined

SECONDARY OUTCOMES:
Effects of H4 deep rTMS on cannabis use frequency | End of intervention period (~4 weeks) and 1-month follow-up
  Cannabis use frequency, as measured by percentage of cannabis use days in the past 7 days.
Effects of H4 deep rTMS on Cannabis craving | End of intervention period (~4 weeks) and 1-month follow-up
  Cannabis cravings will be measured by the Marijuana Craving Scale (12-item scale, higher scores indicate more cravings).
Effects of H4 deep rTMS on motivation to quit Cannabis | End of intervention period (~4 weeks) and 1-month follow-up
  Motivation to quit Cannabis use will be measured by the Readiness Ruler (0-10 scale), higher scores indicate more motivation to quit.
Effects of H4 deep rTMS on resting state neural activity | End of intervention period (~4 weeks) and 1-month follow-up
  Resting state electroencephalography (EEG) will be assessed to examine neural activity changes in the brain.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data and supporting documents will be made available following the publication of the primary findings.
Access Criteria: Doctoral-level researcher with an appointment at professional research organization.